CLINICAL TRIAL: NCT05446727
Title: Quadratus Lumborum Block Versus Erector Spinal Block - Comparison of the Effectiveness of the Analgesic Effect in Patients After Abdominal Surgery
Brief Title: Quadratus Lumborum Block vs Erector Spinal Block for Post Abdomen Surgery Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072.6120.32.2022
Record Dates: First submitted 2022-06-02; First posted 2022-07-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2023-06

CONDITIONS: Pain, Acute; Postoperative Pain; Anesthetics, Local
Keywords: Anesthetics; Local Anesthetics
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus Lumborum block group (Experimental): Experimental: Quadratus Lumborum block group Patients were placed in the lateral decubitus position. After skin disinfection, a linear high-frequency ultrasound probe guarded with a sterile cover was set above the iliac crest and shifted cranially until the three abdominal wall muscles were distinguished. Then, it was moved medially until latissimus dorsi and quadratus lumborum (QLM) muscles were shown within identical short-axis views. A 21-gauge needle was inserted from the edge of the probe using an in-plane technique and advanced into the fascia over the QLM. After ensuring negative aspiration for blood, 30 ml of 0.35% ropivacaine bilateral was injected slowly into the fascial interspace.
  Interventions: Drug: Ropivacaine injection
- erector spinae planae block (Experimental): The ESP block was performed with the patient in a sitting position. After skin disinfection, a linear high-frequency (L14-6NS) ultrasound probe, covered with a sterile sheath, was positioned sagittally 1-2 cm lateral to the midline at the level of the ninth thoracic vertebra (T9). The T9 level was earlier identified by palpating the spinous process of the seventh cervical vertebra and counting down nine intervertebral spaces. After identifying the erector spinae muscle (ESM) and transverse process, a 21-gauge needle was inserted deep into the ESM in a cranio-caudal direction, using an in-plane technique. The needle was advanced, ensuring that it crossed all muscle layers until it contacted the transverse process. A total of 60 mL of 0.35% ropivacaine was given. This procedure was performed bilaterally on each patient.
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — 30ml of 0.35% ropivacaine bilaterally

SUMMARY:
Prior to surgery, patients will be stratified into groups according to the type of surgical procedure. The anticipated groups are as follows:

Patients with colorectal cancer

Patients with prostate cancer

Patients with renal cancer

Patients undergoing surgery for gallbladder cholelithiasis. The Erector Spinal Block (ESP) is based on the deposition of the local anesthetic in the inter-fascial space between the dorsal extensor muscle and the intercostal muscles at the height of the transverse processes. The scope of the blockade covers the dorsal and ventral branches of the thoracic spinal nerves, but also in most cases the investigetors are able to obtain a wide distribution of the drug into the paravertebral space by "permeating" the local anesthetic through the fascial compartments. The clinical effect of the blockade is due to blocking the nerve structures of the paravertebral space (spinal nerve branches and the sympathetic trunk). The scope of the blockade, after its execution at the level of Th5, most often includes the segments from Th1 to L1.

Currently, the Quadratus Lumborum block (QL block) is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery. The local anesthetic injected via the approach of the anterior QL block ( QL1 block ) can more easily extend beyond the TAP to the thoracic paravertebral space or the thoracolumbar plane, the posterior QL block entails a broader sensory-level analgesic and may generate analgesia from T7 to L1.

DETAILED DESCRIPTION:
In abdomen surgery, overall pain is a conglomerate of three different and clinically separate components: incisional pain (somatic pain), visceral pain (deep intra abdominal pain), and shoulder pain due to peritoneal stretching and diaphragmatic irritation associated with carbon dioxide insufflation. Moreover, it has been hypothesized that intense acute pain after labdomen surgery may predict development of chronic pain. Without effective treatment, this ongoing pain may delay recovery, mandate inpatient admission, and thereby increase the cost of such care.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring abdomen surgery
* Patients of age 18 and over
* BMI < 40
* Patients who are expected to stay in-hospital overnight after surgery

Exclusion Criteria:

* Patient refusal
* Contraindications to paravertebral blocks: Infection at the site of needle insertion, empyema, allergy to local anesthetic drugs, and tumor occupying the thoracic paravertebral space, coagulopathy, bleeding disorder or therapeutic anticoagulation
* Known allergy to local anesthetics
* Inability to provide informed consent
* Inability to use a PCA due to languate or comprehension barriers
* BMI >= 40
* Any patient on opioids for greater than or equal to 3 months duration prior to surgery
* Patients with chronic pain syndromes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Total long acting opioid consumption in oxycodone equivalents | 1 days
  the total dosage of given drug

SECONDARY OUTCOMES:
Pain scores will be recorded at intervals. The Numerical Rating Scale (NRS) is an 11-point scale where 0 is no pain and 10 is the worst pain imaginable. | 1 days
  The patients will be asked about level of pain every 2 hours
Incidence of postoperative nausea-vomiting; itching; local anesthetic toxicity; | 1vdays
  The patients will be asked about Incidence of postoperative nausea-vomiting; itching; local anesthetic toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University, Krakow, Maloposkie, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomasz S, Pawel M, Michal C, Szpunar W, Jan S, Tomasz L, Anna K, Renata B, Olga S, Tomasz D, Michal T. Effects of Erector Spinae Plane Block and Quadratus Lumborum Block on Postoperative Opioid Consumption in Laparoscopic Kidney Surgery: A Randomized Controlled Clinical Trial. Pain Res Manag. 2025 Aug 4;2025:8869716. doi: 10.1155/prm/8869716. eCollection 2025. PMID 40791636